CLINICAL TRIAL: NCT01366326
Title: A Multiple-Dose, Open-Label Study to Evaluate the Pharmacokinetics of MNTX in Healthy Adult Subjects
Brief Title: Evaluate the Pharmacokinetics (PK) of Methylnaltrexone (MNTX) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1109
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Methylnaltrexone bromide
  Interventions: Drug: Methylnaltrexone bromide

INTERVENTIONS:
Drug: Methylnaltrexone bromide — Subcutaneous MNTX

SUMMARY:
MNTX 1109 is a single center, open label study, composed of normal healthy adult subjects to evaluate the PK of MNTX and its metabolites administered once daily as a subcutaneous (SC) injection for a period of seven days. Blood samples will be obtained at screening and for drug concentration data.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight ≥40 kg (88 lb)
2. In good health with no clinically significant abnormal findings on the physical examination, medical history or the screening 12-lead ECG
3. Non-smoker
4. Has no known allergies to study drug or other related chemically-related compounds (i.e. naltrexone, naloxone).

Exclusion Criteria:

1. History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease
2. History of clinically significant allergies
3. Positive urine screen for drugs
4. History of positive blood screen for human immunodeficiency virus (HIV), hepatitis B virus (Hep B), or hepatitis C virus (HCV)
5. Prior exposure, allergy or known hypersensitivity to methylnaltrexone
6. Diagnosis of alcohol or substance dependence within the past 12 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of MNTX and its Metabolites | 7 days
  To evaluate the PK profile of MNTX and its metabolites when administered as a SC injection once daily for seven days in healthy adult subjects.

SECONDARY OUTCOMES:
Peak Time of Maximum Concentration (Tmax) of MNTX and its Metabolites | 7 Days
  To evaluate the PK profile of MNTX and its metabolites when administered as a SC injection once daily for seven days in healthy adult subjects.
Area Under the Plasma Concentration versus Time Curve (AUC) of MNTX and its Metabolites. | 7 Days
  To evaluate the PK profile of MNTX and its metabolites when administered as a SC injection once daily for seven days in healthy adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States